CLINICAL TRIAL: NCT03457779
Title: Pilot Study To Investigate Targetable Metabolic Pathways Sustaining Triple Negative (TN) Breast Cancer and Associated Genomic Alterations
Brief Title: Pilot Study To Investigate Targetable Metabolic Pathways Sustaining Triple Negative Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 017-396
Record Dates: First submitted 2018-02-08; First posted 2018-03-08 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Glucose

STUDY DESIGN:
Intervention Model Description: Patients with TNBC will receive [1,2-13C]-glucose IV to prior to undergoing a biopsy of their breast cancer and blood collection to allow for in depth evaluation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Non Glucose Arm (Experimental): 4 patients without glucose infusion
  Interventions: Dietary Supplement: Glucose
- Glucose Arm (Experimental): 12 Patients with glucose infusion
  Interventions: Dietary Supplement: Glucose

INTERVENTIONS:
Dietary Supplement: Glucose — The first 4 patients enrolled on trial will undergo the research core biopsies of their TNBC without the 13C glucose infusion; these samples will serve as control tissue that will be processed identically to the tissues obtained from patients who received the glucose isotope.
  The following 12 patients will receive 6 grams (g) of [1,2-13C] glucose as an IV

SUMMARY:
The primary objective is to describe and discover new insights into the glucose, amino acid, and lipid metabolic dependencies of TNBC via nuclear magnetic resonance (NMR) spectroscopy analysis of in vivo [1,2-13C] glucose-labeled breast cancer biopsies.

The secondary objectives are to correlate the dominant metabolic dependencies of TNBCs with pathologic response to preoperative chemotherapy, and with the cancers' molecular signaling pathways assessed via NGS and RPPA.

DETAILED DESCRIPTION:
One of the recognized hallmarks of cancer cells is deregulated cellular metabolism, characterized by enhanced metabolic autonomy compare with non-transformed cells. Tumor cells typically display an overall increase in glucose metabolism, associated with enhanced aerobic glycolysis and decreased oxidative phosphorylation, accompanied by a requirement for a high rate of protein, nucleotide, and fatty acid synthesis to provide the raw materials for cell division. 13C-glucose is a non-radioactive stable isotope tracer that has been widely used in vitro, in vivo, and in patients in a variety of disease settings to study glucose, amino acid, and lipid metabolism, at steady state and following intervention. [1,2-13C] glucose can provide additional information on the activity of the oxidative pentose phosphate pathway versus glycolysis. Administration of intravenous 13C-glucose is a convenient and affordable approach to analyzing the metabolomics of human cancers in their native microenvironments.

The metabolic dependencies of the various breast cancer subtypes are poorly understood. Importantly, in depth analyses of the in situ metabolic processes utilized by triple-negative breast cancers (TNBCs) using state-of-the-art in vivo [1,2-13C]-glucose infusions in patients with TNBC has never been done. In TNBC, oncogenic activation of key signaling pathways leads to altered metabolic programming resulting in an increased dependence on exogenous nutrients such as glucose and glutamine. These data further suggest a hypothesis that TNBCs may employ a cellular mechanism called macropinocytosis to ingest and degrade interstitial albumin to accumulate glutamine. This process may then be exploited for therapeutic gain through enhanced uptake by cells that utilize macropinocytosis to meet their metabolic requirements.

In this study, administration of [1,2-13C]-glucose to patients with TNBC will be done prior to patients undergoing a biopsy of their breast cancer as well as blood sample collection which will allow for in depth evaluation of glycolysis as well as lipid and amino acid metabolism by Joshua Rabinowitz, PhD, at Princeton University who is an international expert in cancer metabolomics. RAS and PI3K pathway and other genomic alterations as well as pathway activation status will be determined by next generation sequencing (NGS) and by reverse phase protein array (RPPA), and will be correlated with the metabolic findings, and both will be assessed in the context of the patients' response to standard preoperative chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

A patient will be considered for enrollment in this study if all the following criteria are met:

1. Female patients ≥18 years of age.
2. Have TNBC defined as invasive ductal cancer: ER- tumors with <10% of tumor nuclei immunoreactive; PR- tumors with <10% of tumor nuclei immunoreactive; HER2-negative defined as follows:

   1. FISH-negative (FISH ratio <2.0), or
   2. IHC 0-1+, or
   3. IHC 2+ AND FISH-negative (FISH ratio<2.0)
3. Adequate hematologic function, defined by:

   1. Absolute neutrophil count (ANC) >1000/mm3
   2. Platelet count ≥100,000/mm3
   3. Hemoglobin >9 g/dL (in the absence of red blood cell transfusion)
4. Adequate liver function, defined by:

   1. AST and ALT ≤ 5 x the upper limit of normal (ULN)
   2. Total bilirubin ≤1.5 x ULN
5. Adequate renal function, defined by:

   a. Serum creatinine ≤ 2 x ULN or calculated creatinine clearance of ≥60 ml/min
6. Have blood glucose <250 mg/dL
7. Willing to undergo 1 mandatory core biopsy (6 passes) for research purposes.
8. All patients must be able to understand the investigational nature of the study and give written informed consent prior to study entry.

Exclusion Criteria:

A patient will be ineligible for inclusion in this study any of the following criteria are met:

1. Patients receiving any anti-cancer therapy (chemotherapy, immunotherapy, and/or biologic therapy).
2. Is currently enrolled, or will enroll in, a different clinical study in which investigational therapeutic procedures are performed or investigational therapies are administered while participating in this study.
3. Has a history of insulin-dependent diabetes.
4. Concomitant active malignancy
5. Is pregnant or breastfeeding.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients ≥18 years of age.
Enrollment: 16 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2020-04-08 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Amount of glucose, amino acid, and lipid metabolites in TNBC. | 2 years
  Amount of glucose, amino acid, lipid will be measured in 16 patients with TNBC using NMR spectroscopy to see how metabolism is affected in TNBC.

SECONDARY OUTCOMES:
Correlation of signaling pathways in TNBC with response and metabolites. | 2 years
  A panel of key cancer cell signaling pathways will be analyzed in TNBC tissues from 16 patients using phosphoproteomic technology and next generation sequencing. The activated and deactivated pathways will be correlated with standard of care pathologic response (residual disease or no residual disease) and amount of glucose, amino acid, and lipid metabolized.

CONTACTS AND LOCATIONS:
Overall Officials: Joyce O'Shaughnessy, MD, Principal Investigator — Texas Oncology/Baylor Scott & White Health
Locations (1):
- Baylor University Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
For serum collection and storage at the Baylor BPM core, until they are shipped to Princeton University. The key metabolic dependency findings will be correlated with genomic and proteomic alterations assessed by NGS and RPPA, and with patients' response to preoperative chemotherapy.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be shared from opening of recruitment through study closure.
Access Criteria: De-Identified Data will be shared via encrypted email

REFERENCES:
- [Derived] Ghergurovich JM, Lang JD, Levin MK, Briones N, Facista SJ, Mueller C, Cowan AJ, McBride MJ, Rodriguez ESR, Killian A, Dao T, Lamont J, Barron A, Su X, Hendricks WPD, Espina V, Von Hoff DD, O'Shaughnessy J, Rabinowitz JD. Local production of lactate, ribose phosphate, and amino acids within human triple-negative breast cancer. Med. 2021 Jun 11;2(6):736-754. doi: 10.1016/j.medj.2021.03.009. Epub 2021 Apr 14. PMID 34223403